CLINICAL TRIAL: NCT05754619
Title: Le Emozioni Negli Stili di Comunicazione e Relazione di Genitori Con Figli Emofilici.
Brief Title: Emotions in the Communication and Relationship Styles of Parents With Hemophilic Children.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, De Cristofaro Raimondo, Prof. Raimondo De Cristofaro, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 4913
Record Dates: First submitted 2023-02-03; First posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-02

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 7 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with HA: 20 parents with hemophilic children. The sample will consist of 10 mothers and 10 fathers.

SUMMARY:
Severe hemophilia is a rare, inherited, X-linked disorder. Currently, standard therapy involves ev infusion of drugs from a very young age.

The diagnosis of hemophilia is a traumatic event for the parents, even before the unborn child. The management of the hemophilia patient involves the whole family. Also in relation to its heredity.Focus on the ways in which parents of children with hemophilia manage their emotional experience.

DETAILED DESCRIPTION:
Severe hemophilia is a rare, inherited, X-linked disorder. Currently, standard therapy involves ev infusion of drugs from a very young age.The diagnosis of hemophilia is a traumatic event for the parents, even before the unborn child. The management of the hemophilia patient involves the whole family. Also in relation to its heredity.Focus on the ways in which parents of children with hemophilia manage their emotional experience.he diagnosis of hemophilia brings with it, in parents, fears, guilt, overprotective temptations that push us to act rather than to narrate the meaning of that need of ours, caregiving modes that risk engaging our operational side at the expense of recognizing ourselves and our feelings and emotions. We have no reason to think that that traumatic stimulus installs in us an atypical mode of resorting to our emotional intelligence. Therefore, it becomes even more significant to study parent-child communication processes on this target, to observe whether and how the adult's emotional area finds its place and expression. On the results of this work, the foundations could be laid for subsequent observational or interventional studies.

ELIGIBILITY:
Inclusion Criteria:

* Haemophilia A

Exclusion Criteria:

* No Informed Conset

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: the study includes 20 caregivers, parents of childrens (10-18 yo) with Haemophilia
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-10-14 (Actual); Primary Completion 2023-05-14 (Estimated); Study Completion 2023-05-14 (Estimated)

PRIMARY OUTCOMES:
The study aims to highlight the ways in which the caregivers of haemophiliac children and young people manage and express their emotional experience through interviews and reports | 1 month
  The study aims to highlight the ways in which care givers of hemophilic children and youth manage and express their emotional experiences. It therefore intends to answer these questions:
  * How do parents of hemophilic children and youth contribute to the development of their children's emotional intelligence?
  * What adult role model do they consciously or unconsciously propose in relation to frailties and fears?
  * How do they guide their children in dealing with frailties and fears?
  * Does the communication process they construct integrate their experience and is it congruent with it?

SECONDARY OUTCOMES:
opportunity for mirroring the parents interviewed by which they construct participation in their child's life in the experience of illness with interview and questionnaire. | 3 months
  This study represents a potential opportunity for mirroring the interviewed parents, who in nonjudgmental observation will be able to see themselves and the unconscious dynamics by which they construct participation in their child's life in the experience of illness. Where interviewed parents show willingness and interest, a thirty-minute follow-up meeting will be held fifteen days/one month later, which will aim to accommodate their experience following the stimuli offered by the experience with our team. The main purpose, then, is in accompanying these people to process what will have emerged in the interview-interview

CONTACTS AND LOCATIONS:
Overall Officials: Raimondo De Cristofaro, MD, Principal Investigator — Fondazione Policlinico Universitario A.Gemelli IRCCS Rome
Locations (1):
- FPG, Roma, Italy